CLINICAL TRIAL: NCT02836977
Title: Maintenance Tegafur-uracil Versus Observation Following Adjuvant Oxaliplatin-based Regimen in Patients With Stage III Colon Cancer After Radical Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20160016
Record Dates: First submitted 2016-07-10; First posted 2016-07-19 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-06

CONDITIONS: Stage III Colon Cancer
Keywords: tegafur-uracil
MeSH Terms: conditions — Colonic Neoplasms | interventions — Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- maintenance therapy (Experimental): Patients will receive oral tegafur-uracil 400mg/day (100mg/Cap., 2 capsules each time, twice a day), combined with oral folinic acid 30mg/day (15mg/Tab., 1 tablet each time, twice a day), and continue for one year.
  Interventions: Drug: tegafur-uracil
- observation arm (Active Comparator): Patients will be observed following adjuvant oxaliplatin-based regimen.
  Interventions: Drug: tegafur-uracil

INTERVENTIONS:
Drug: tegafur-uracil — Eligible patients will receive tegafur-uracil orally at a dose of 400mg/day (100mg/Cap., 2 capsules each time, twice a day) and folinic acid 30mg/day (15mg/Tab., 1 tablet each time, twice a day) for one year.
  Other Names: UFUR

SUMMARY:
Primary Objective:

To compare 3-year disease free survival (DFS) of tegafur-uracil following adjuvant oxaliplatin-based regimen to observation following adjuvant oxaliplatin-based regimen in patients with stage III colon cancer after radical resection.

Secondary Objectives:

* To assess 5-year overall survival (OS) in each arm
* To assess the safety profiles

DETAILED DESCRIPTION:
Objectives:

1. Primary Objective:

   To compare 3-year disease free survival (DFS) of tegafur-uracil following adjuvant oxaliplatin-based regimen to observation following adjuvant oxaliplatin-based regimen in patients with stage III colon cancer after radical resection.
2. Secondary Objectives:

   * To assess 5-year overall survival (OS) in each arm
   * To assess the safety profiles

Patient Selection and Enrollment:

Number of Subjects: Eligible patients will be randomized in 2 arms in the ratio of 2:1, to reach approximately 546 patients in total.

Plan of the Study:

1. Study Design This is an open-label, randomized, comparative, double arm, multicenter study to assess disease free survival, overall survival, safety profiles with tegafur-uracil following adjuvant oxaliplatin-based regimen as maintenance for one-year in patients with stage III colon cancer after radical resection in Taiwan.
2. Subject Number Eligible patients will be randomized in 2 arms in the ratio of 2:1, to reach approximately 546 patients in total.
3. Study Schedule Study date: the time getting approval letter issued by both regulatory authority and institutional review board (IRB) Expected recruitment rate: 23 subjects/month Duration of recruitment: at least 2 years. Duration of the study: at least 5 years.
4. Visit Schedule The schedule of assessments (please refer section 8.4 for the details) indicates the number and timing of the planned visits, which must be maintained as accurately as possible. The visit schedule must be maintained as accurate as possible.
5. Duration of Treatment Treatment should be administered up to maximum one year, disease progression, intolerable toxicity, or consent withdrawal during any time of the study, the patient will be withdraw.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each subject must fulfill all of the following criteria:

1. pathologically confirmed colon carcinoma;
2. stage III disease (T1-4, N1-2, M0 as defined by AJCC 7th Edi.);
3. completion of adjuvant oxaliplatin-based regimen without evidence of any recurrent disease;
4. entry of the trial within 3 weeks after adjuvant oxaliplatin-based regimen;
5. performance status of ECOG 0, 1, 2;
6. age between 20 and 80 years old;
7. written informed consent to participate in the trial.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded from the trial:

1. previous or current systemic malignancy with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ, unless there has been a disease-free interval of at least 5 years;
2. inadequate hematopoietic function defined as below:

   1. hemoglobin < 9 g/dL;
   2. absolute neutrophil count (ANC) < 1,500/mm3;
   3. platelet count < 100,000/mm3;
3. inadequate organ functions defined as below:

   1. total bilirubin > 2 times upper limit of normal (ULN);
   2. hepatic transaminases (ALT and AST) > 2.5 x ULN;
   3. creatinine > 1.5 x ULN;
4. other significant medical conditions that are contraindicated to tegafur-uracil or render patient at high risk from treatment complications based on investigator's discretion;
5. presence of other serious concomitant illness;
6. participation in another clinical trial with any investigational drug within 30 days prior to entry;
7. pregnant or lactating women or women of childbearing potential.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | three to six months

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yeh YS, Tsai HL, Huang CW, Wei PL, Sung YC, Tang HC, Wang JY. Maintenance tegafur-uracil versus observation following an adjuvant oxaliplatin-based regimen in patients with stage III colon cancer after radical resection: study protocol for a randomized controlled trial. Trials. 2017 Apr 26;18(1):191. doi: 10.1186/s13063-017-1904-9. PMID 28441966